CLINICAL TRIAL: NCT01281085
Title: Validation of a Kinematic Functional Shoulder Score Including Only Essential Movements: a Pilot Study
Brief Title: Validation of a Score for Shoulder Function Evaluation Based on Movement Analysis
Status: Completed | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: Réseau d'études appliquées des pratiques de Santé de Réadapation (ré)insertion (Unknown)
Responsible Party: Claude Pichonnaz, HES professor, HECVSanté, filière physiothérapie
Other Study IDs: SAGEX-24519
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Shoulder Pain
Keywords: Shoulder; Outcome treatment; Validation Studies; Biomechanics
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Shoulder conditions including rotator cuff condition treated conservatively, shoulder instability treated conservatively, diaphyseal humerus fracture or subcapital humerus fracture treated surgically and frozen shoulder

SUMMARY:
Questionnaires are frequently used to evaluate shoulder function in various diseases or after surgery. However, measurement of shoulder function is presently a controversial issue. Shoulder movement analysis based on embedded sensors could be a promising alternative to questionnaires. Some studies already demonstrated the relevance of this approach. It has also been demonstrated that a simple testing procedure including only two arm movements produces comparable results to more complicated testing procedures. However, more studies are needed to extensively establish if this simplified testing procedure provides a trustworthy evaluation of patient shoulder function and its evolution.

This study is a preliminary study which aims to develop a precise testing procedure which will be used in a future study aiming to evaluate measurement properties of a simple shoulder function test based on movement sensors.

DETAILED DESCRIPTION:
Background Measurement of shoulder function is a controversial issue. There is a great variety of measurement tools but none of them has been universally accepted. There is therefore a need to develop extensively validated and convenient measurement tools.

Embedded computerized movement analysis can potentially meet these requirements for measurement of shoulder function. Ambulatory measurement devices allow application in various clinical conditions, display adequate precision and accuracy, and are considerably more straightforward than laboratory-based systems.

Using a Physilog ® II embedded system, Coley (2007) developed a relatively simple score of shoulder function (P Score). The method is based on arm power measurement by three-dimensional accelerometers and gyroscopes during seven consecutive shoulder movements. It demonstrated reliability, responsiveness and criterion-based validity. However, additional knowledge and technological progress could now contribute to further simplification of the.

A secondary analysis of Coley's study data based on principal component analysis and multiple regressions highlighted that a procedure including only two selected movements produces comparable results to P Score. Moreover, the development of wireless systems considerably simplifies set up. Consequently, simpler but equivalent measurement procedure can now be considered.

However some important issues have to be clarified before an extensive validation study can be undertaken. The simplicity of the testing procedure allows test replication. However, the number of movement replications needed to obtain a reliable outcome is presently unknown. Relevance of testing procedure and study feasibility have also to be evaluated. A pilot study is needed to clarify these issues.

Aim The aim of this pilot study is to determine the number of movement replications needed to obtain a reliable result using a simplified cinematic shoulder measurement procedure as well as to evaluate testing procedure and study protocol.

Methods Measurement will be carried out with four groups of patients presenting with frequent shoulder conditions (rotator cuff condition, shoulder instability, diaphyseal or subcapital humerus fracture, frozen shoulder). Measurement procedure includes two consecutive measurements, alternatively conducted by two evaluators. Currently used functional questionnaires will be completed at both stages.

Statistical analysis will address outcome variability according to number of replications and reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff condition, conservative treatment indicated
* Shoulder instability, conservative treatment indicated
* Diaphyseal humerus fracture or subcapital humerus fracture treated surgically, at 6 weeks post surgery
* Frozen shoulder, conservative treatment indicated

Exclusion Criteria:

* Bilateral shoulder condition or other shoulder condition than the ones mentioned in inclusion criteria
* Any concomitant pain or condition involving upper limb
* Cervical spine condition involving upper limb pain or mobility restriction
* Insufficient French language level to understand patient information form, consent form or questionnaires
* Insufficient ability to give truly informed consent or to understand questionnaires. It will be proceeded to a Mini Mental State score in case of uncertainty, with exclusion criteria at 24 points/30 (ANAES 2000).
* Medical contraindication to execute movements required for score completion
* Tumor
* Neurological condition interfering with test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a shoudler condition, as stated during the medical examination performed at the specialized shoulder consultation of the hospital
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
variability of kinematic simplified functional score | only one measurement session
  This pilot study mainly aims at defining how many tests replications are needed to obtain a reliable shoulder function measurement

SECONDARY OUTCOMES:
intra- and inter-reproducibility of kinematic functional shoulder score | only one measurement session
  As measurement are performed twice respectively by two evaluators, this pilot study will provide a first insight of test reliability

CONTACTS AND LOCATIONS:
Overall Officials: Claude A. Pichonnaz, PT MSc, Principal Investigator — HECVSanté and CHUV-UNIL
Locations (1):
- Département de l'Appareil Locomoteur - CHUV, Lausanne, Switzerland

REFERENCES:
- [Background] Coley B, Jolles BM, Farron A, Bourgeois A, Nussbaumer F, Pichonnaz C, Aminian K. Outcome evaluation in shoulder surgery using 3D kinematics sensors. Gait Posture. 2007 Apr;25(4):523-32. doi: 10.1016/j.gaitpost.2006.06.016. Epub 2006 Aug 28. PMID 16934979